CLINICAL TRIAL: NCT04492462
Title: The Impact of Two Different Physical Therapy Programs in the Rehabilitation of Patients Undergoing Anterior Approach Hip Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Stephen Kayiaros MD, Principal Investigator, Clinical Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro20140001090
Record Dates: First submitted 2020-06-29; First posted 2020-07-30 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Hip Arthritis; Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Anterior Approach; Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formal Physical Therapy (Experimental)
  Interventions: Other: Formal Physical Therapy
- Self-directed Physical Therapy (Experimental)
  Interventions: Other: Self-directed Physical Therapy

INTERVENTIONS:
Other: Formal Physical Therapy — Patients will undergo standard physical therapy following their surgery with a physical therapist in an office
  Arms: Formal Physical Therapy
Other: Self-directed Physical Therapy — Patients will undergo self-directed physical therapy in the comfort of their own home by completing a list of exercises and stretches without the direct supervision of a physical therapist in a physical therapist office
  Arms: Self-directed Physical Therapy

SUMMARY:
This study will look to determine two different types of physical therapy regimens in patients who undergo anterior total hip replacement. We will compare the results of two groups. The first group, the "Formal Physical Therapy" group, will undergo standard physical therapy following their surgery. They will see a physical therapist in a physical therapy office after their surgery. Here, the therapist will work with the patient to strengthen muscles and improve their walking. The second group, the "Self-directed Physical Therapy" group, will undergo physical therapy in the comfort of their own home using common household items (chairs, steps, etc). These patients will be given a list of exercises and stretches to perform on their own. It is our goal to prove that formal physical therapy is not needed after anterior hip replacements.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years of age
* Patients undergoing primary anterior total hip arthroplasty for the diagnosis of osteoarthritis
* Patients with no previous invasive hip surgery (such as a previous hip replacement)

Exclusion Criteria:

* Non-English speaking persons will be excluded in our study.
* Patients with a recent history (<1 year) of heart attack, stroke, and lung clots.
* Previous invasive surgery on the hip undergoing replacement
* Patients with dementia, Parkinson's, or other neurological disorders
* Non-ambulatory patients
* Patients with impaired ability to consent, whether because of mental illness or otherwise
* Patients being discharged to a rehabilitation center
* Patients that experience intra-operative complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change inHarris Hip Score (HHS) | assessed 1,3,6, and 12 months after total hip replacement to assess change at each time point following surgery
  elf-administered health survey that assesses pain, function, absence of deformity, and range of motion of the hip through 10 questions. HHS measures dysfunction, so a higher score indicates a better, higher functional outcome. Less than 70 is poor result, 70-80 ia fair result, 80-90 is good result, 90-100 is excellent result

SECONDARY OUTCOMES:
Change in timed up and go test | assessed 1,3,6, and 12 months after total hip replacement to assess change at each time point following surgery
  Patients will be assessed the amount of time it takes for them rise from a standard arm chair, walk 10 feet on the floor at normal pace, and then return and site down in same standard arm chair. Duration to complete task will be recorded in seconds
Change in Visual Analog Scale for Pain | assessed 1,3,6, and 12 months after total hip replacement to assess change at each time point following surgery
  Patients will rate their pain on a scale form 0-10 at a given time point with 0 being no pain and 10 being unbearable pain. The higher the number, the more pain
Change in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) form | assessed 1,3,6, and 12 months after total hip replacement to assess change at each time point following surgery
  Self-administered health survey that assesses pain, stiffness, and function of arthritis of the hip or knee. WOMAC form assesses activities of daily living, functional mobility, gait, general health, pain, and quality of life. WOMAC questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). A total score of 0 to 96 is possible, with a lower score indicating less pain or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Kayiaros, MD, Principal Investigator — Rutgers University
Locations (2):
- United States (2):
  - University Orthopaedic Associates, Somerset, New Jersey
  - Robert Wood Johnson Somerset Hospital, Somerville, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR